CLINICAL TRIAL: NCT02623803
Title: Perioperative Intravenous Lidocaine Infusion for Patients Undergoing Laparoscopic and Open Pancreatectomies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elird Bojaxhi, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-003955
Record Dates: First submitted 2015-11-16; First posted 2015-12-08 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pancreatectomy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): lidocaine infusion will be initiated at the time of anesthesia induction in the operating room. Dosage 1.5mg/kg/hour. Continuous infusion until patient meets discharge criteria in recovery room.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): placebo infusion (D5W) will be initiated at the time of anesthesia induction in the operating room. Continuous infusion until patient meets discharge criteria in recovery room.
  Interventions: Drug: Placebo D5W

INTERVENTIONS:
Drug: Lidocaine
  Arms: Treatment group
Drug: Placebo D5W
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate if a lidocaine infusion will provide benefit to pancreatectomy patients in regards to analgesia and return of bowel function.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing elective open or laparoscopic total pancreatectomies and pancreatoduodenectomies (i.e., Whipple procedure), and participating in the Enhanced Recovery Protocol (ERP) at Mayo Clinic in Florida.
* Age 18 - 80 years old
* American Society of Anesthesiologist (ASA) class I - III
* BMI < 40
* Ability to understand and read English

Exclusion Criteria:

* Not able or willing to sign consent
* Intolerance or allergy to opioids, NSAIDS, acetaminophen, or amide-type local anesthetics (i.e., lidocaine).
* History of epilepsy or currently receiving treatment for seizures
* Severe hepatic insufficiency (Child-Pugh Score C)
* Renal insufficiency (creatinine clearance less than 30 mL/minute)
* Advance heart failure (NY Heart failure stage 3 or greater; Ejection function <30%)
* Cardiac arrhythmias: 2nd and 3rd degree heart block, sick sinus syndrome, symptomatic bradyarrhythmias, Wolff-Parkinson-White (WPW) syndrome, or Stokes-Adams syndrome; Left bundle branch block or bifascicular block; Not to exclude patients the following conditions unless clinical circumstance dictate: Atrial fibrillation or atrial fluTter; Presence of Implantable Cardioverter Defibrillator (ICD), or pacemakers
* Patients on anti-arrhythmic therapy (i.e., digoxin, amiodarone, flecainide, lidocaine, sotalol, etc.). Not to exclude patients on beta blockers (i.e., metoprolol, atenolol, etc.) unless clinical circumstance dictate
* Patients with active psychiatric disorders or cognitive dysfunction
* Pregnancy or lactating
* Enucleation, central, and distal pancreatectomy
* Opioid tolerance (defined as consumption of greater than 30 mg of oxycodone per day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elird Bojaxhi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] DE CLIVE-LOWE SG, DESMOND J, NORTH J. Intravenous lignocaine anaesthesia. Anaesthesia. 1958 Apr;13(2):138-46. doi: 10.1111/j.1365-2044.1958.tb08045.x. No abstract available. PMID 13521304
- [Background] BARTLETT EE, HUTSERANI O. Xylocaine for the relief of postoperative pain. Anesth Analg. 1961 May-Jun;40:296-304. No abstract available. PMID 14448503
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Wallin G, Cassuto J, Hogstrom S, Linden I, Faxen A, Rimback G, Hedner T. Effects of lidocaine infusion on the sympathetic response to abdominal surgery. Anesth Analg. 1987 Oct;66(10):1008-13. PMID 3631561
- [Background] Wheatley RG, Schug SA, Watson D. Safety and efficacy of postoperative epidural analgesia. Br J Anaesth. 2001 Jul;87(1):47-61. doi: 10.1093/bja/87.1.47. No abstract available. PMID 11460813
- [Background] Senagore AJ, Delaney CP, Mekhail N, Dugan A, Fazio VW. Randomized clinical trial comparing epidural anaesthesia and patient-controlled analgesia after laparoscopic segmental colectomy. Br J Surg. 2003 Oct;90(10):1195-9. doi: 10.1002/bjs.4223. PMID 14515286
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Herroeder S, Pecher S, Schonherr ME, Kaulitz G, Hahnenkamp K, Friess H, Bottiger BW, Bauer H, Dijkgraaf MG, Durieux ME, Hollmann MW. Systemic lidocaine shortens length of hospital stay after colorectal surgery: a double-blinded, randomized, placebo-controlled trial. Ann Surg. 2007 Aug;246(2):192-200. doi: 10.1097/SLA.0b013e31805dac11. PMID 17667496
- [Background] Rimback G, Cassuto J, Tollesson PO. Treatment of postoperative paralytic ileus by intravenous lidocaine infusion. Anesth Analg. 1990 Apr;70(4):414-9. PMID 2316883
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Gower ST, Quigg CA, Hunt JO, Wallace SK, Myles PS. A comparison of patient self-administered and investigator-administered measurement of quality of recovery using the QoR-40. Anaesth Intensive Care. 2006 Oct;34(5):634-8. doi: 10.1177/0310057X0603400514. PMID 17061640
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: lidocaine infusion will be initiated at the time of anesthesia induction in the operating room. Dosage 1.5mg/kg/hour. Continuous infusion until patient meets discharge criteria in recovery room.
  Lidocaine
- Control Group: placebo infusion (D5W) will be initiated at the time of anesthesia induction in the operating room. Continuous infusion until patient meets discharge criteria in recovery room.
  Placebo D5W
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 25 | 23
Completed | 25 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.5) | 65.1 (13.3) | 65.7 (67.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 15 | 9 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (4.2) | 28.0 (5.4) | 27.1 (4.8)
American Society of Anesthesiologists (ASA) Physical Status Classification [Count of Participants; unit: Participants] — Measure Description: ASA classification defines ASA I as a normal healthy patient, ASA II as a patient with a mild systemic disease without substantive functional limitations and an ASA III as a patient with a severe systemic disease with substantive functional limitations. A lower classification (I/II) is a more positive reflection of overall health compared to a higher classification (III).
  Participants
    ASA II | 3 | 6 | 9
    ASA III | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Pain in Postoperative Period
Description: Overall pain will be measured upon arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: baseline - arrival at the PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 20 | 18
score on a scale | 1.6 (3.2) | 2.7 (1.0)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.1459, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Opioid Consumption
Description: Total opioid consumption in PACU converted to morphine equivalents in mg.
Time Frame: up to 4 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 23 | 18
mg | 3.9 (4.1) | 6.7 (7.6)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.2050, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain at Rest
Description: Pain will be measured at rest upon arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: baseline - arrival at the PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 23
score on a scale | 2.1 (3.6) | 2.6 (3.3)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.3989, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain With Coughing
Description: Pain with coughing will be measured upon arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: baseline - arrival at the PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 15
score on a scale | 2.3 (3.9) | 2.5 (3.2)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.5285, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Overall Pain
Description: Overall pain will be measured 30 minutes after arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 30 minutes after arrival to PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 19 | 18
score on a scale | 3.3 (3.1) | 5.3 (3.3)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.0697, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Pain at Rest
Description: Pain at rest will be measured 30 minutes after arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 30 minutes after arrival to PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 22
score on a scale | 3.3 (3.6) | 5.1 (3.6)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.1029, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Pain With Coughing
Description: Pain with coughing will be measured 30 minutes after arrival at the post-operative care unit (PACU) using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 30 minutes after arrival to PACU
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 19 | 16
score on a scale | 4.3 (3.9) | 5.8 (3.1)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.3136, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Overall Pain
Description: Overall pain will be measured approximately 12 hours post-operatively using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: approximately 12 hours post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 22 | 17
score on a scale | 4.4 (2.7) | 5.4 (2.8)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.2196, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pain at Rest
Description: Pain at rest will be measured approximately 12 hours post-operatively using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: approximately 12 hours post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 20
score on a scale | 4.0 (3.0) | 5.0 (3.2)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.3057, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Pain With Coughing
Description: Pain with coughing will be measured approximately 12 hours post-operatively using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: approximately 12 hours post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 13 | 9
score on a scale | 4.7 (3.1) | 7.6 (2.4)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.0404, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Overall Pain
Description: Overall pain will be measured on post-operative day 1 at 1am using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1am
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale | 5.1 (2.0) | 5.5 (2.1)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.5314, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Pain at Rest
Description: Pain at rest will be measured on post-operative day 1 at 1 am using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1 am
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 23
score on a scale | 4.0 (3.1) | 4.6 (1.9)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.3166, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Pain With Coughing
Description: Pain with coughing will be measured on post-operative day 1 at 1 am using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1 am
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 9
score on a scale | 5.4 (3.4) | 7.1 (2.1)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.2363, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Overall Pain
Description: Overall pain will be measured on post-operative day 1 at 1 pm using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1 pm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 20 | 18
score on a scale | 4.8 (1.8) | 4.8 (1.8)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.9171, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Pain at Rest
Description: Pain at rest will be measured at post-operative day 1 at 1 pm using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1 pm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 24 | 22
score on a scale | 4.0 (2.3) | 4.8 (2.4)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.4194, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Pain With Coughing
Description: Pain with coughing will be measured on post-operative day 1 at 1 pm using numerical rating scale (NSR). Subjects will rate their pain after surgery on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: post-operative day 1 at 1 pm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 8
score on a scale | 5.4 (2.7) | 5.8 (3.1)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.7073, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Length of Time to First Flatus
Description: Time of first instance of flatus will be measured as the number of days post operatively for bowel function to return.
Time Frame: up to 3 weeks postoperatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 23 | 23
days | 3.9 (6.6) | 2.7 (1.2)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.5107, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Length of Time to First Bowel Movement
Description: Time of first instance of a bowel movement will be measured as the number of days post operatively for bowel function to return.
Time Frame: up to 3 weeks postoperatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 18 | 18
days | 5.8 (7.7) | 5.2 (6.0)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.8339, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Total Opioid Consumption
Description: Total amount of opioids converted to morphine equivalents in mg administered in the first 24 hours after surgery.
Time Frame: up to 24 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 25 | 23
mg | 7.4 (5.4) | 7.9 (6.4)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.8927, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Quality of Recovery
Description: This questionnaire is a short 15 question form that measures the quality of a subject's postoperative recovery. The scale is ranked from 0 to 10, where 0 is a poor response and 10 is an excellent response.
Time Frame: Day 15 post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 20 | 21
score on a scale
  Able to breathe easily | 9.1 (1.8) | 8.7 (1.8)
  Been able to enjoy food | 6.2 (3.7) | 5.4 (2.9)
  Feeling rested | 7.2 (1.8) | 6.0 (2.2)
  Have had a good sleep | 7.1 (1.9) | 6.6 (2.4)
  Able to look after personal toliet and hygiene | 9.2 (2.3) | 8.8 (2.3)
  Able to communicate with family or friends | 9.6 (1.1) | 9.3 (1.4)
  Getting support from hospital doctors and nurse | 8.8 (3.1) | 9.5 (0.7)
  Able to return to work or usual home activities | 5.4 (3.5) | 4.9 (3.2)
  Feeling comfortable and in control | 7.1 (2.5) | 6.7 (2.7)
  Having a feeling of general well-being | 7.5 (2.2) | 6.7 (2.2)
  Moderate pain | 7.9 (2.5) | 6.6 (2.7)
  Severe pain | 9.4 (1.8) | 8.8 (2.2)
  Nausea or vomiting | 8.6 (2.3) | 8.2 (2.6)
  Feeling worried or anxious | 7.7 (3.0) | 7.6 (2.5)
  Feeling sad or depressed | 8.4 (2.6) | 7.8 (3.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time patient initiated study drug infusion until hospital discharge (approximately 5-7 days).
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02623803/Prot_SAP_000.pdf